CLINICAL TRIAL: NCT02482285
Title: Assessment of Frailty in Elderly Patients With Advanced Cancers
Acronym: FAC-C
Status: Terminated | Type: Observational
Why Stopped: Difficulty recruiting. Study aims now overlap standard of care assessments and future planned studies.
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 6731
Record Dates: First submitted 2015-06-12; First posted 2015-06-26 (Estimated); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and baseline, week 12 and weeks 24
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is looking at the feasibility of performing frailty assessments on elderly patients with advanced cancers

DETAILED DESCRIPTION:
This study is primarily looking to see if it is feasible to assess frailty in patients age 70 years and above with advanced cancers. it is also evaluating whether there may be any correlation between these assessments and toxicity and treatment and outcome.

The assessments include: Frailty score, nutritional assessment, comorbidity score and quality of life. In addition sarcopenia will be assessed using timed walk, grip strength and muscle mass measurement from imaging performed as part of routine clinical care.

The assessments will be performed at baseline, week 12 and week 24.

There is the option for patients to also donate blood samples for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of advanced carcinoma - not suitable for curative treatment
* Age 70 years or over
* seen by an oncologist for consideration of palliative systemic medical therapy and decision regarding management already made
* WHO Performance Status 0-2
* Written informed consent

Exclusion Criteria:

* Hepatocellular cancer
* Prostate cancer
* Breast cancer

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with advanced cancers
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2014-06-04 (Actual); Primary Completion 2016-01-25 (Actual); Study Completion 2016-01-25 (Actual)

PRIMARY OUTCOMES:
Percentage patients consenting for assessments out of number approached | Baseline
  Number of patients consenting for the study as a percentage of number of patients approached about the study.
Time taken to complete assessments | Baseline, week 12 and week 24
  Length of time participants take to complete study assessments

SECONDARY OUTCOMES:
Frailty as a predictor of grade 3/4 toxicity | baseline
  Evaluate whether there is a possible correlation between frailty score at baseline and development of grade 3/4 toxicity during anticancer treatment
Sarcopenia as a predictor of outcome | baseline, week 12 and week 24
  sarcopenia at baseline and over time as a predictor of outcome
Quality of life EORTC QCQ 30 | baseline, week 12 and week 24
  Participants complete EORTC QCQ 30 questionnaire
Biomarker assessment of frailty and associated factors which may include genetic analysis | baseline, week 12 and week 24
  Assessment of frailty biomarkers in blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Alastair Greystoke, MRCP, PhD, MBChB, MSc, Principal Investigator — Newcastle University
Locations (1):
- Newcastle upon Tyne NHS Trust, Newcastle upon Tyne, United Kingdom